CLINICAL TRIAL: NCT05481242
Title: An Observational Study About Adverse Outcomes in Acute Pulmonary Embolism Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YIZHUO GAO, Doctor, Shengjing Hospital
Other Study IDs: AOAPE
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism and Thrombosis; Deterioration, Clinical
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective observational study — retrospective observational study

SUMMARY:
This multi-center retrospective study collected clinical, laboratory, and CT pulmonary angiography parameters with acute pulmonary embolism patients from admission to predict adverse outcomes within 30 days after admission into hospital.

DETAILED DESCRIPTION:
This multi-center retrospective study collected clinical, laboratory, and CT pulmonary angiography parameters with acute pulmonary embolism patients from admission to predict adverse outcomes within 30 days after admission into hospital.

Eligible patients were collected to develop and evaluate a simple predictive model for predicting the adverse outcomes. The discriminatory power was evaluated by comparing the nomogram to the established risk stratification systems. The consistency of the nomogram was evaluated using the validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 18 years and a pulmonary embolism diagnosis based on CT pulmonary angiography

Exclusion Criteria:

* pregnancy
* reception of reperfusion treatment before admission
* missing data regarding CT parameters, echocardiography, cardiac troponin I (c-Tn I), and N-terminal-pro brain natriuretic peptide (NT-pro BNP) levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse outcomes | 30 days
  The endpoints of deterioration in this study were defined as the occurrence of any adverse clinical outcomes from medical records and follow-up within 30 days of admission such as death, mechanical ventilation, cardiopulmonary resuscitation, and the need for life-saving vasopressor or reperfusion treatment .In each centre, the researchers for evaluating endpoints were blind to collect and to measure study parameters.

SECONDARY OUTCOMES:
Adverse outcomes | 2 years
  The endpoints of deterioration in this study were defined as the occurrence of any adverse clinical outcomes from medical records and follow-up within 2 years of admission such as death, mechanical ventilation, cardiopulmonary resuscitation, and the need for life-saving vasopressor or reperfusion treatment .In each centre, the researchers for evaluating endpoints were blind to collect and to measure study parameters.

CONTACTS AND LOCATIONS:
Overall Officials: DONG JIA, Principal Investigator — Shenjing Hospital of CHINA MEDICAL UNIVERSITY
Locations (1):
- Shenjing Hospital of CHINA MEDICAL UNIVERSITY, Shenyang, Liaoning, China